CLINICAL TRIAL: NCT01141075
Title: A Phase 2 Study of Ataluren (PTC124®) as an Oral Treatment for Nonsense Mutation Methylmalonic Acidemia
Brief Title: Ataluren for Nonsense Mutation Methylmalonic Acidemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low enrollment and unclear pharmacologic effect in available pharmacodynamic data (not due to any safety concerns).
Sponsor: PTC Therapeutics (Industry)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC124-GD-012-MMA
Record Dates: First submitted 2010-06-07; First posted 2010-06-10 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Amino Acid Metabolism, Inborn Errors
MeSH Terms: conditions — Amino Acid Metabolism, Inborn Errors | interventions — ataluren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ataluren (Experimental): Cycle 1: Ataluren treatment will be taken 3 times per day with meals for 28 days at doses of 5 mg/kg (morning), 5 mg/kg (midday), and 10 mg/kg (evening); there will then be an interval of 21 up to 42 days without treatment.
  Cycle 2: Ataluren treatment will be taken 3 times per day with meals for 28 days at doses of 10 mg/kg (morning), 10 mg/kg (midday), and 20 mg/kg (evening); there will then be an interval of 14 days without treatment.
  Interventions: Drug: Ataluren

INTERVENTIONS:
Drug: Ataluren — Ataluren will be provided as a vanilla-flavored powder to be mixed with water.
  Other Names: PTC124

SUMMARY:
Methylmalonic acidemia (MMA) is a rare genetic disorder caused by mutations in the gene for mitochondrial enzyme methylmalonyl-CoA mutase (MCM) or in one of the genes for adenosylcobalamin (AdoCbl). Lack of these proteins causes toxic elevations of methylmalonic acid (MMacid) in blood, urine, and other tissues. A specific type of mutation, called a nonsense (premature stop codon) mutation, is the cause of the disease in approximately 5% to 20% of participants with mutations in the MCM gene, and approximately 20% to >50% of participants with mutations in one of the AdoCbl genes. Ataluren is an orally delivered, investigational drug that acts to overcome the effects of the premature stop codon, potentially enabling the production of functional MCM/AdoCbl. This study is a Phase 2a trial evaluating the safety and activity of ataluren in participants with MMA due to a nonsense mutation. The main purpose of this study is to understand whether ataluren can safely decrease MMacid levels.

DETAILED DESCRIPTION:
In this study, participants with MMA due to a nonsense mutation will be administered an investigational drug called ataluren. Evaluation procedures to determine if a participant qualifies for the study will be performed within 14 days prior to the start of drug administration. Eligible participants who elect to enroll in the study will then participate in 2 drug administration and follow-up periods. Within the first period, ataluren will be taken 3 times per day with meals for 28 days at doses of 5 milligrams/kilograms (mg/kg) (morning), 5 mg/kg (midday), and 10 mg/kg (evening); there will then be an interval of approximately 21 days without ataluren. Within the second period, ataluren will be taken 3 times per day with meals for 28 days at doses of 10 mg/kg (morning), 10 mg/kg (midday), and 20 mg/kg (evening); there will then be an interval of approximately 14 days without ataluren. During the study, ataluren activity, safety, and pharmacokinetics will be evaluated, and MMacid levels in blood and urine will be measured periodically.

ELIGIBILITY:
Major Inclusion Criteria:

* Ability to provide written informed consent (parental/guardian consent if applicable)/assent (if applicable)
* Age ≥2 years
* Phenotypic evidence of methylmalonic acidemia (MMA) based on the presence of characteristic clinical symptoms or signs and an elevated plasma MMacid level (>0.27 micromole/liter (umol/L)
* Presence of a nonsense mutation in at least 1 allele of the mutase (mut), Cobalamin A (cblA), or Cobalamin B (cblB) gene
* Glomerular filtration rate ≥30 milliliters (mL)/minutes/1.73 meters squared (m^2), serum aminotransferase values ≤2.5*the upper limit of normal, serum bilirubin ≤1.5*the upper limit of normal, plasma adrenocorticotropic (ACTH) within normal limits
* Willingness and ability to comply with scheduled visits, drug administration plan, study restrictions, and study procedures

Major Exclusion Criteria:

* Known hypersensitivity to any of the ingredients or excipients of the study drug
* Any change in chronic treatment for MMA within 2 months prior to start of screening laboratory assessments
* Episode of metabolic decompensation within 1 month prior to start of Screening laboratory assessments
* History of organ transplantation
* Ongoing dialysis for renal dysfunction

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07-19 (Actual); Primary Completion 2011-11-03 (Actual); Study Completion 2011-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Barth, MD, Study Director — PTC Therapeutics
Locations (9):
- ZNA Queen Paola Child Hospital and Provincial Centre for Metabolic Disorders, Antwerp, Belgium
- France (2):
  - Hôpital Edouard Herriot, Lyon
  - Necker-Enfants Malades Hospital, Paris
- University Children's Hospital, Düsseldorf, Germany
- Italy (3):
  - Istituti Clinici di Perfezionamento, Milano, Milan
  - Federico II University, Naples
  - University Hospital, Department of Pediatrics, Padua
- University Children's Hospital, Zurich, Switzerland
- Great Ormand Street Hospital, London, United Kingdom

REFERENCES:
- [Background] Welch EM, Barton ER, Zhuo J, Tomizawa Y, Friesen WJ, Trifillis P, Paushkin S, Patel M, Trotta CR, Hwang S, Wilde RG, Karp G, Takasugi J, Chen G, Jones S, Ren H, Moon YC, Corson D, Turpoff AA, Campbell JA, Conn MM, Khan A, Almstead NG, Hedrick J, Mollin A, Risher N, Weetall M, Yeh S, Branstrom AA, Colacino JM, Babiak J, Ju WD, Hirawat S, Northcutt VJ, Miller LL, Spatrick P, He F, Kawana M, Feng H, Jacobson A, Peltz SW, Sweeney HL. PTC124 targets genetic disorders caused by nonsense mutations. Nature. 2007 May 3;447(7140):87-91. doi: 10.1038/nature05756. Epub 2007 Apr 22. PMID 17450125
- [Background] Hirawat S, Welch EM, Elfring GL, Northcutt VJ, Paushkin S, Hwang S, Leonard EM, Almstead NG, Ju W, Peltz SW, Miller LL. Safety, tolerability, and pharmacokinetics of PTC124, a nonaminoglycoside nonsense mutation suppressor, following single- and multiple-dose administration to healthy male and female adult volunteers. J Clin Pharmacol. 2007 Apr;47(4):430-44. doi: 10.1177/0091270006297140. PMID 17389552
- See also: PTC Therapeutics' website — http://www.ptcbio.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Ataluren: Cycle 1: Ataluren treatment was taken 3 times per day with meals for 28 days at doses of 5 milligrams/kilograms (mg/kg) (morning), 5 mg/kg (midday), and 10 mg/kg (evening); there was then an interval of 21 up to 42 days without treatment.
  Cycle 2: Ataluren treatment was taken 3 times per day with meals for 28 days at doses of 10 mg/kg (morning), 10 mg/kg (midday), and 20 mg/kg (evening); there was then an interval of 14 days without treatment.
Period: Cycle 1
Arm/Group | Ataluren
Started | 11
Received at Least 1 Dose of Study Drug | 11
Completed | 11
Not Completed | 0
Period: Cycle 2
Arm/Group | Ataluren
Started | 11
Received at Least 1 Dose of Study Drug | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- Ataluren: Cycle 1: Ataluren treatment was taken 3 times per day with meals for 28 days at doses of 5 mg/kg (morning), 5 mg/kg (midday), and 10 mg/kg (evening); there was then an interval of 21 up to 42 days without treatment.
  Cycle 2: Ataluren treatment was taken 3 times per day with meals for 28 days at doses of 10 mg/kg (morning), 10 mg/kg (midday), and 20 mg/kg (evening); there was then an interval of 14 days without treatment.
Arm/Group | Ataluren
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 12 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Plasma Methylmalonic Acid (MMacid) Levels
Description: Normal plasma MMacid level is <0.27 micromole/liters (umol/L). Plasma samples for MMacid levels were collected after a 2- to 4-hour fast. Plasma MMacid levels were measured by a standard gas chromatography/mass spectroscopy (GC/MS) stable-isotope dilution method. Individual participant values in plasma MMacid levels at Baseline and end-to-treatment (Day 28 and Day 29 [last day of dosing]) in each cycle were recorded.
Time Frame: Baseline and Day 28 and Day 29 (last day of dosing) of Cycles 1 and 2
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: umol/L
Arm/Group | Ataluren
Number analyzed (Participants) | 11
umol/L
  Baseline of Cycle 1 | 153.7 [15.5 to 971.5]
  Day 28 of Cycle 1 | 160.3 [20.5 to 1163.3]
  Day 29 of Cycle 1 | 175.9 [20.4 to 1432.9]
  Baseline of Cycle 2 | 196.5 [29.3 to 933.1]
  Day 28 of Cycle 2 | 280.9 [22.8 to 1083.3]
  Day 29 of Cycle 2 | 188.1 [20.7 to 1390.4]

2. Secondary Outcome: Urinary MMacid Levels
Description: The normal urinary MMacid level is <4 millimole/mole (mmol/mol) creatinine. Urinary samples for MMacid levels were collected after a 2- to 4-hour fast. Urinary MMacid levels were measured by a standard GC/MS stable-isotope dilution method.
Time Frame: Baseline and Day 28 and Day 29 (last day of dosing) of Cycles 1 and 2
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: mmol/mol creatinine
Arm/Group | Ataluren
Number analyzed (Participants) | 11
mmol/mol creatinine
  Baseline of Cycle 1 | 1870.8 [84.9 to 10875.7]
  Day 28 of Cycle 1 | 1953.0 [100.9 to 12768.5]
  Day 29 of Cycle 1 | 1364.6 [173.2 to 31412.4]
  Baseline of Cycle 2 | 1577.7 [241.8 to 16603.9]
  Day 28 of Cycle 2 | 1479.1 [162.6 to 8914.4]
  Day 29 of Cycle 2 | 1588.3 [150.1 to 14063.2]

3. Secondary Outcome: Plasma Propionylcarnitine Levels
Description: Plasma samples for propionylcarnitine levels were evaluated to detect disease activity. The level of propionylcarnitine was measured using gas chromatography and LC/MS-MS. An increase in propionylcarnitine values indicates greater disease activity.
Time Frame: Baseline and Day 28 and Day 29 (last day of dosing) of Cycles 1 and 2
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: umol/L
Arm/Group | Ataluren
Number analyzed (Participants) | 11
umol/L
  Baseline of Cycle 1 | 7.5 [1.8 to 39.1]
  Day 28 of Cycle 1 | 6.9 [2.2 to 17.6]
  Day 29 of Cycle 1 | 4.3 [1.9 to 16.8]
  Baseline of Cycle 2 | 6.6 [1.0 to 33.9]
  Day 28 of Cycle 2 | 5.5 [0.9 to 19.6]
  Day 29 of Cycle 2 | 4.5 [0.4 to 17.6]

4. Secondary Outcome: Urine Methylcitric Acid Levels
Description: Urine methylcitric acid levels were evaluated to detect disease activity. An increase in methylcitric acid values indicates greater disease activity.
Time Frame: Baseline and Day 28 and Day 29 (last day of dosing) of Cycles 1 and 2
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Median (Full Range); unit: mmol/mol creatinine
Arm/Group | Ataluren
Number analyzed (Participants) | 11
mmol/mol creatinine
  Baseline of Cycle 1 | 48.1 [10.2 to 309.5]
  Day 28 of Cycle 1 | 124.2 [12.0 to 380.3]
  Day 29 of Cycle 1 | 83.2 [17.3 to 498.4]
  Baseline of Cycle 2 | 84.9 [14.2 to 211.0]
  Day 28 of Cycle 2 | 72.3 [35.7 to 243.5]
  Day 29 of Cycle 2 | 65.1 [30.3 to 201.3]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the Investigator on a scale of mild, moderate and severe, with severe as an AE that prevents usual activities. Relationship of AE to treatment was determined by the Investigator. Serious AEs include death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized the participant and required medical intervention to prevent the previously listed serious outcomes. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Day 112 (end of study follow-up)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 11
Participants
  Any AE | 10
  Severe AE | 0
  Treatment-related AE | 3
  Serious AE | 0
  AE leading to discontinuation | 0

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Laboratory (Hematology and Biochemistry) Abnormal Results
Description: Hematological and biochemistry data graded according to Common Terminology Criteria for Adverse Events (CTCAE) severity grade (Grade 1 [mild], Grade 2 [moderate], Grade 3 [severe], Grade 4 [life-threatening], or Grade 5 [fatal]). Life-threatening (Grade 4) or severe (Grade 3) laboratory abnormalities were considered clinically significant. Recurrent or persistent moderate (Grade 2) abnormalities were also considered clinically significant in certain circumstances. Hematology assessments: white blood cell count with differential, hemoglobin, hematocrit, other red cell parameters, and platelet count. Biochemistry assessments: sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, magnesium, calcium, phosphorus, uric acid, glucose, total protein, albumin, bilirubin (direct and indirect), aspartate aminotransferase, alanine aminotransferase, glutamyl transferase, creatine kinase, lactate dehydrogenase, alkaline phosphatase, total cholesterol, and triglycerides.
Time Frame: Baseline up to Day 112 (end of study follow-up)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 11
Participants
  With at least 1 hematology abnormality | 0
  With at least 1 biochemistry abnormality | 2

7. Secondary Outcome: Number of Participants With a Metabolic Decompensation Episode
Description: A metabolic decompensation episode is characterized by vomiting, hypotonia, and alteration of consciousness associated with metabolic acidosis and hyperammonemia.
Time Frame: Baseline up to Day 112 (end of study follow-up)
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 11
Participants | 0

8. Secondary Outcome: Number of Participants Compliant With Study Treatment
Description: For each participant, compliance was described in terms of the proportion of drug actually taken relative to the amount that should have been taken during the time the participant was on study (both Cycle 1 and Cycle 2).
Time Frame: Baseline up to Day 29 of Cycles 1 and 2
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Ataluren
Number analyzed (Participants) | 11
Participants
  Received all doses of study drug | 11
  Received at least 1 different dose than planned | 4

9. Secondary Outcome: Ataluren Plasma Exposure
Description: Validated quantitative methods employing high performance liquid chromatography with tandem mass spectroscopy (HPLC-MS-MS) were used to determine plasma concentrations of unchanged ataluren. The median and full range of the total of all of the ataluren plasma concentrations collected at Baseline and at Day 28 are reported.
Time Frame: Baseline on Day 0 of Cycles 1 and 2 [0 (predose), 1, 2, 3, and 4 hours postdose of the morning dose and 0 (predose) of the midday dose]; Day 28 of Cycles 1 and 2 [0 (predose), 1, 2, 3, and 4 hours postdose of the morning, midday, and evening doses]
Population: All randomized participants who received at least 1 dose of study drug and had evaluable ataluren plasma exposure data.
Measure: Median (Full Range); unit: microgram/milliliters (μg/mL)
Arm/Group | Ataluren
Number analyzed (Participants) | 11
microgram/milliliters (μg/mL)
  Baseline of Cycle 1: number analyzed (Participants) | 7
  Baseline of Cycle 1 | 6.1 [1.3 to 16.3]
  Day 28 of Cycle 1: number analyzed (Participants) | 9
  Day 28 of Cycle 1 | 6.6 [0.6 to 29.9]
  Baseline of Cycle 2: number analyzed (Participants) | 10
  Baseline of Cycle 2 | 14.5 [3.2 to 29.2]
  Day 28 of Cycle 2: number analyzed (Participants) | 9
  Day 28 of Cycle 2 | 13.2 [1.8 to 44.8]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 112 (end of study follow-up)
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Ataluren
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 10/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ataluren (N=11)
Glomerular vascular disorder (Renal and urinary disorders) | 2
Hypercreatininaemia (Renal and urinary disorders) | 2
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Haematoma (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Muscle strain (Injury, poisoning and procedural complications) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Convulsion (Nervous system disorders) | 1
Nasopharyngitis (Infections and infestations) | 4
Pyrexia (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Headache (Nervous system disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review.

The sponsor may consult with the PI to require changes to the communication or extend the embargo.